CLINICAL TRIAL: NCT04183712
Title: A Multicentre, Open-label, Randomised, Controlled Study of Target Therapy Based on Tumor Molecular Profiling With GEMOX in Recectable Gallbladder Carcinoma Patients Monitored by ctDNA.
Brief Title: Target Therapy With GEMOX in Recectable Gallbladder Carcinoma Patients Monitored by ctDNA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Ruijin Hospital (Other); RenJi Hospital (Other); Qilu Hospital of Shandong University (Other); The First Affiliated Hospital of Anhui Medical University (Other); Shanghai East Hospital of Tongji University (Other); Changshu Affiliated Hospital of Soochow University (Other); Qinghai People's Hospital (Other); The Second People's Hospital of Baoshan, Yunnan Province (Unknown); Lanzhou University Second Hospital (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); The First People's Hospital of Nantong (Unknown)
Responsible Party: Principal Investigator, Yingbin Liu, MD, PhD, FACS, Prof., Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LTGBCLYB2019
Record Dates: First submitted 2019-11-28; First posted 2019-12-03 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Gallbladder Carcinoma
MeSH Terms: conditions — Gallbladder Neoplasms | interventions — Gemcitabine; Oxaliplatin; Commerce; Long-Term Synaptic Depression; Afatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Afatinib with GEMOX (Experimental): Patients will receive targeted therapy(Afatinib 40mg orally from day 1 to day 21 combined with GEMOX chemotherapy(gemcitabine 1000 mg/m2 on days 1 and 8 of each cycle by IV infusion and oxaliplatin 100 mg/m2 on day 1 of each cycle by IV infusion)
  Interventions: Drug: gemcitabine and oxaliplatin.; Drug: Afatinib
- GEMOX (Active Comparator): Patients will receive conventional GEMOX chemotherapy (gemcitabine 1000 mg/m2 on days 1 and 8 of each cycle by IV infusion and oxaliplatin 100 mg/m2 on day 1 of each cycle by IV infusion）
  Interventions: Drug: gemcitabine and oxaliplatin.

INTERVENTIONS:
Drug: gemcitabine and oxaliplatin. — GEMOX Conventional chemotherapy:gemcitabine and oxaliplatin.
  Other Names: Gemzar(Eli Lilly and Company) and Aiheng(Jiangsu Hengrui Medicine Co., Ltd.)
Drug: Afatinib — Target therapy Drug: afatinib
  Other Names: Gilotrif(Boehringer-Ingelheim)
  Arms: Afatinib with GEMOX

SUMMARY:
The purpose of this study is to evaluate the feasibility, efficacy and safety of target therapy according to genomic and proteomic profiling combined with GEMOX in recectable gallbladder carcinoma patients monitored by ctDNA.

DETAILED DESCRIPTION:
Genomic profiling studies the deoxyribonucleic acid (DNA) of a tumor to detect genetic changes or abnormalities. immuno-histochemistry tests reveal the abnormal activation status of signal pathways involved in study. These information will be used to recommend target therapy which may be more likely to result in a beneficial response. Patients will receive target antitumor agents according to the result of genomic and proteomic profiling and be monitored by circulating tumor DNA(ctDNA).

ELIGIBILITY:
Inclusion Criteria:

* Chinese#
* Stable vital signs, ECOG:0-1;
* Patients have a diagnosis of resectable gallbladder carcinoma by histopathology or cytopathology after radical surgery.
* Adequate fresh tumor tissue for genome sequencing and immunohistochemistry test; harboring mutations or abnormal activation of erb-b2 receptor tyrosine kinase signal pathway components
* Life expectancy of more than 18 weeks;
* T stage≥ T2 or histopathological lymph node positive according to AJCC (8th edition) staging.
* Adequate hepatic, hematologic and renal functions(ALT≤5×upper limit of normal (ULN), AST≤5×ULN, the Child-Pugh classification for class A or B, white blood cells≥3×10^9/L, neutrophils≥1.5×10^9/L, platelets≥75×10^9/L , hemoglobin ≥ 90g/L, creatinine clearance rate≥60ml/min;
* Volunteer for this study, have written informed consent and have good Patient compliance;
* Female patients of childbearing potential and their mates agree to avoid pregnancy.

Exclusion Criteria:

* Have received following treatment before this study: a. Anti-tumor molecular target therapy; anti-tumor chemotherapy in 6 months; b. lesions have been treated by irradiation; c. participate in other therapeutic or interventional clinical trials.
* History of other malignancies except carcinoma in-situ of uterine cervix, cured basal cell carcinoma of skin and other malignancies for more than 5 years;
* Have serious concurrent illness including, but not limited to uncontrolled congestive heart failure(NYHA classification grade III or IV), unstable angina pectoris, unstable cardiac arrhythmias, uncontrolled moderate or serious hypertension(systolic blood pressure >21.3 Kpa or diastolic blood pressure >13.3 Kpa);
* Have ongoing or active serious infection;
* Have uncontrolled diabetes mellitus;
* Psychiatric illness which potentially hamper the ability to willingly give written informed consent and compliance with the study protocol;
* Active autoimmune diseases require long-term use of steroids or received allotransplantation
* Other serious illness considered not suitable for this study by investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
3-year DFS | up to 3 years
  3-year disease free survival rates:The progression is defined consistent with contrast enhanced MRI/CT.

SECONDARY OUTCOMES:
3-year OS | up to 3 years
  3-year Overall survival rates

OTHER OUTCOMES:
sensitivity and specificity of ctDNA | up to 2 years
  sensitivity and specificity of ctDNA compared to clinical index（CA199，CEA）for monitoring tumour progression

CONTACTS AND LOCATIONS:
Overall Officials: Yingbin Liu, PHD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (2):
- China (2):
  - Renji hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang M, Zhao Y, Li Y, Cui X, Liu F, Wu W, Wang XA, Li M, Liu Y, Liu Y. Afatinib in combination with GEMOX chemotherapy as the adjuvant treatment in patients with ErbB pathway mutated, resectable gallbladder cancer: study protocol for a ctDNA-based, multicentre, open-label, randomised, controlled, phase II trial. BMJ Open. 2023 Feb 28;13(2):e061892. doi: 10.1136/bmjopen-2022-061892. PMID 36854604